CLINICAL TRIAL: NCT07355361
Title: Multicenter, Randomized, Parallel-Controlled Clinical Trial on Huaier Granule for Proteinuria Associated With Immunotherapy and Anti-Angiogenic Therapy in Breast Cancer Patients
Brief Title: Huaier Granule and Proteinuria
Acronym: N093
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of Breast Surgery Department, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N093
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Proteinuria; Breast Cancer Patients
Keywords: proteinuria; Immunotherapy; Anti-angiogenic therapy; Breast cancer patients
MeSH Terms: conditions — Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Group (Active Comparator): Antitumor therapy + Proteinuria management + Huaier Granule treatment
  Interventions: Drug: Huaier Granule; Drug: Antitumor therapy; Drug: Proteinuria Management
- B Group (Active Comparator): Proteinuria management + Huaier Granule treatment
  Interventions: Drug: Antitumor therapy; Drug: Proteinuria Management

INTERVENTIONS:
Drug: Huaier Granule — Huaier Granule Group: Participants will take Huaier Granule (Z20000109) on top of their standard treatment. The dosing is 10g, orally, three times a day. Treatment continues until the study ends, or an event such as disease progression, unacceptable side effects, withdrawal, or death occurs, whichever comes first. The investigator can also stop treatment if it's no longer deemed beneficial. Refer to the drug label for details. The investigator will decide on continued use if the background cancer therapy is changed due to progression.
  Arms: A Group
Drug: Antitumor therapy — The pre-existing regimen started before enrollment, subject to adjustment based on clinical routine.
Drug: Proteinuria Management — Specialist-managed care (including follow-up or drug therapy [excluding Huaier Granule]) initiated post-proteinuria diagnosis.

SUMMARY:
The goal of this clinical trial is to learn if adding Huaier Granule to standard care can treat proteinuria (excess protein in the urine) in adult female breast cancer patients (aged 18-75) who developed this condition as a side effect of their immunotherapy or anti-angiogenic cancer treatment.

The main question it aims to answer is:

* Does the addition of Huaier Granule to standard care improve the effectiveness of proteinuria treatment after 8 weeks?

Researchers will compare the group receiving standard care plus Huaier Granule to the group receiving standard care alone to see if the combination is more effective at reducing protein levels in the urine.

Participants will:

* Be randomly assigned to one of the two study groups.
* Continue their prescribed anti-cancer therapy (immunotherapy or anti-angiogenic therapy).
* Receive standard medical care for proteinuria from a kidney specialist.
* If in the experimental group, take Huaier Granule orally, three times a day.
* Attend clinic visits every 4 weeks for up to 24 weeks for check-ups and tests, including urine and blood tests.

ELIGIBILITY:
Inclusion Criteria:

* **Inclusion Criteria**

  1. Female patients aged 18-75 years.
  2. Histopathologically confirmed diagnosis of breast cancer.
  3. Currently receiving or having a prior history of immunotherapy and/or anti-angiogenic therapy.
  4. First-time detection of proteinuria on urinalysis, graded as +, ++, or +++.
  5. 24-hour urinary protein quantification between 0.15g and 3.5g (exclusive).
  6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
  7. Karnofsky Performance Status (KPS) score ≥70.
  8. No prior treatment with Huaier Granule within one month before enrollment.
  9. Life expectancy of at least 6 months.
  10. Willingness to voluntarily participate in the study and provision of signed informed consent.

Exclusion Criteria:

* **Exclusion Criteria**

  1. Known history of chronic kidney disease (eGFR <60 ml/min/1.73m²) or diabetic nephropathy.
  2. Proteinuria attributed to other diseases, including but not limited to primary renal disease, hypertension, urinary tract infection, systemic lupus erythematosus, or multiple myeloma.
  3. Current use of ACEI/ARB medications (unless the dosage has been stable for ≥4 weeks prior to enrollment).
  4. Known allergy, contraindication, or specific precaution to any component of Huaier Granule.
  5. Women who are pregnant, breastfeeding, or planning to conceive.
  6. Concurrent participation in any other clinical trial investigating medications for proteinuria.
  7. Any other condition that, in the judgment of the investigator, would make the patient unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Response rate of proteinuria treatment at Week 8 | From enrollment to the end of treatment at 8 weeks.
  The proportion of subjects (across both groups) achieving a best overall response of Complete Response, Partial Response, or Stable Disease in proteinuria at 8 weeks.

SECONDARY OUTCOMES:
Response rate of proteinuria treatment at Week 16 | From enrollment to the end of treatment at 16 weeks
  Response rate at Week 16 (defined as the proportion of subjects with complete response, partial response, or stable disease in proteinuria)
Change from baseline in 24-hour urinary protein quantification at Weeks 8 and 16 | From enrollment to the end of treatment at 16 weeks
  The between-group difference in the mean change from baseline in 24-hour urinary protein quantification at Week 8.
Mean percent reduction in 24-hour urinary protein quantification at Weeks 8 and 16 | From enrollment to the end of treatment at 16 weeks
  The mean of the percentage change, which is calculated for each subject as: (Baseline 24-hour urinary protein value - Week 8 value) / Baseline value × 100%, averaged across all subjects in both the experimental and control groups.
Other Renal Adverse Events at Weeks 8 and 16 | From enrollment to the end of treatment at 16 weeks
  The incidence and severity of other renal adverse events (including but not limited to elevated blood pressure, increased serum creatinine, elevated blood urea nitrogen, acute kidney injury, nephritis, nephrotic syndrome, and renal failure) are defined as follows:
  Incidence is defined as the proportion of subjects experiencing any of the specified other renal adverse events within the respective total population.
  Severity will be graded according to the criteria described in the section for definitions and assessment of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ming Shao, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided